CLINICAL TRIAL: NCT02808741
Title: F901318 - A Two Part Study Designed to Evaluate the Single and Multiple Dose Pharmacokinetics of an Immediate Release Tablet Formulation of F901318
Brief Title: Evaluation of Immediate Release Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F901318-01-07-16
Record Dates: First submitted 2016-06-11; First posted 2016-06-22 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-06

CONDITIONS: Invasive Aspergillosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- F901318 SDD (Experimental): Liquid formulation
  Interventions: Drug: F901318 SDD
- F901318 IR (Experimental): Solid formulation
  Interventions: Drug: F901318 IR
- F901318 IR Fasting (Experimental): Fasting solid formulation
  Interventions: Drug: F901318 IR Fasting
- F901318 IR Fed (Experimental): Fed solid formulation
  Interventions: Drug: F901318 IR Fed

INTERVENTIONS:
Drug: F901318 SDD — Pharmacokinetics area under curve
  Arms: F901318 SDD
Drug: F901318 IR — Pharmacokinetics area under curve
  Arms: F901318 IR
Drug: F901318 IR Fasting — Pharmacokinetics area under curve
  Arms: F901318 IR Fasting
Drug: F901318 IR Fed — Pharmacokinetics area under curve
  Arms: F901318 IR Fed

SUMMARY:
Single dose comparison of liquid and solid formulation, followed by study of effect of high fat breakfast.

Evaluation of multiple dose pharmacokinetics and tolerability

DETAILED DESCRIPTION:
The study will be split into 2 parts, Part 1, ( A and B), and Part 2.

Part 1A Part 1A of the study will be a single centre, open label, 2-way crossover in healthy male and female volunteers and will assess the relative bioavailability of a single 360 mg dose (as 3 x 120mg tablets) of F901318 IR tablet formulation in comparison to a 360 mg dose of an SDD suspension for oral dosing. It is planned that 10 volunteers will be enrolled to Part 1A of the study. These 10 subjects will continue into Part 1B of the study.

There will be a minimum washout of 10 days between doses provided to volunteers.

Following Part 1A there will be a two week period of interim analysis during which safety and pharmacokinetic data will be reviewed. In order to assess doses within the therapeutic range in Part 1B, a decision will be made using the available data, on whether the dose of F901318 IR tablet formulation should be altered. Dose will be altered by amending the number of units dosed.

Part 1B Following the dose decision meeting where data obtained in Part 1A of the study is reviewed, the selected dose of F901318 IR tablet formulation will be assessed in a further single centre, open label, 2-way crossover in healthy male and female volunteers. The selected dose will be administered in the fed (30 minutes following an FDA high fat meal) and fasted states in a randomised fashion. .

There will be a minimum washout of 10 days between doses provided to volunteers.

Following Part 1B there will period a period of interim analysis during which safety and pharmacokinetic data will be reviewed. In order to assess doses within the therapeutic range in Part 2, a decision will be made using the available data, on the dose of F901318 IR formulation to be dosed in Part 2. Dose will be altered by amending the number of units dosed. It will also be determined if doses in Part 2 will be administered in the fed or fasted state.

Part 2 In part 2, the dose(s) anticipated to yield therapeutic plasma concentrations will be tested over a 10-day period. This will be a double blind placebo controlled, randomised, parallel group design in 10 healthy male and female subjects, 8 taking active compound and 2 taking placebo. In order to mimic the expected treatment schedule in phase 2 trials, it is anticipated that there will be a loading dose given over 1 or 2 days, followed by once daily or twice daily doses of study drug up to a total of 10 days.

In both parts of the study, blood will be drawn for safety and pharmacokinetic evaluation. Adverse events, vital signs and 12 lead ECGs will be monitored throughout. In Part 1, Holter monitoring will be performed for 12 hours after each dose. Part 2, ECG Holter monitoring will be performed on Days 1 and 10 only.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be healthy males or females of any ethnic origin between 18 and 55 years of age and weighing between 50-100 kg (body mass index of 18.0-32.0 kg/m2 inclusive).
2. Females of child bearing potential must be established on a reliable form of contraception and have a negative pregnancy test at screening.
3. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is acceptable).
4. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions.

Exclusion Criteria:

1. Subjects who do not have suitable veins for multiple vene-punctures/cannulation as assessed by the investigator at screening
2. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
3. Male or female subjects who are not willing to use appropriate contraception during the study and until 3 months after the last dose.
4. Subjects who have received any prescribed systemic or topical medication within 14 days of the dose administration unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 120 hours
  Area Under Concentration Time Curve

SECONDARY OUTCOMES:
Treatment emergent adverse events | 120 hours
  Incidence of Treatment-Emergent Adverse Events [Safety]).

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No